CLINICAL TRIAL: NCT06282952
Title: NEwborn Infant of a Mother With Obesity - Fecal Microbiome Transplantation, a Randomized Controlled Trial
Brief Title: NEwborn Infant of a Mother With Obesity - Fecal Microbiome Transplantation, RCT
Acronym: NEMO-FMT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oulu University Hospital (Other)
Collaborators: University of Oulu (Other); University of Turku (Other); Turku University Hospital (Other Government); University of Helsinki (Other); Academy of Finland (Other); Biocenter Oulu (Unknown)
Responsible Party: Principal Investigator, Marika Paalanne, MD, PhD, Associate Professor, Oulu University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 198/2023
Record Dates: First submitted 2023-10-16; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Fecal Microbiota Transplantation; Cesarean Section; Overweight and Obesity
Keywords: Fecal Microbiota Transplantation; Cesarean Section; Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: The eligible women are randomized into two groups in which their newborns receive either fecal microbiota transplant from 1) their own mother (50 newborns) or 2) the Microbiome Biobank (50 newborns). The randomization 1:1 is done in blocks of 4 mothers. The study is double blinded. If mother has Group B streptococcus colonization or other infectious disease described in table 1, and microbiota transplant cannot be given or if mother will have non-elective-CS and the microbiome transplant is not available, the mother is included in 3) the observational cohort, which is "open" (not blinded).
Who Masked: Participant, Care Provider, Investigator
Masking Description: The research statistician performs the computer-generated randomization. The study nurse prepares the fecal transplant according to the randomization. Study participants or investigators are not aware of study group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Fecal microbiota transplant from biobank (Experimental): The newborns receive fecal microbiota transplant from their own mother (50 newborns).
  Interventions: Dietary Supplement: Fecal transplant
- Fecal microbiota transplant from own mother (Active Comparator): Newborns receive fecal microbiota transplant from normal weight, healthy female donor from the Microbiome Biobank (50 newborns).
  Interventions: Dietary Supplement: Fecal transplant
- The observational cohort (No Intervention): If mother has Group B streptococcus (GBS) colonization or other infectious, and microbiota transplant cannot be given or if mother will have non-elective-CS and the microbiome transplant is not available, the mother is included in the observational cohort, which is "open" (not blinded).

INTERVENTIONS:
Dietary Supplement: Fecal transplant — At delivery, the fecal transplant is thawed and 0.5 mL representing 3.5 mg of the mother's or donors' fecal sample is dissolved in 5 mL of the mother's own milk or when not available pasteurized bank milk. The sample is given orally to newborn infants as soon as possible but not later than 6 h of delivery and not later than two hours after defrosting.
  Arms: Fecal microbiota transplant from biobank; Fecal microbiota transplant from own mother

SUMMARY:
The goal of this clinical trial is to investigate the differences in microbiota, height and weight between infants born by cesarean section to obese mothers and randomized to receive fecal microbiota transplant after birth. The main questions it aims to answer are:

* Could fecal transplant be used improve gut microbiota and prevent overweight or obesity.
* Is the source of colonization a modifiable factor and can it be changed by using an early fecal microbiota transplant.

DETAILED DESCRIPTION:
1. BACKGROUND

   In recent decades, the prevalence of obesity in children has increased dramatically worldwide. Obese children and adolescents are around five times more likely to be obese in adulthood than those who are not obese. Although childhood obesity is a complex and multifactorial outcome, it seems that obese children have different gut microbiome already at birth. Many of the previous studies highlight maternal risk factors such as higher maternal BMI before pregnancy, excess gestational weight gain, gestational diabetes (GDM) and C-section as a risk factor for childhood overweight or obesity. Perinatal factors, in particular the birth by Cesarean section as well as perinatal antibiotics, have also been identified as a critical determinant of early-life microbiota composition and development. However, the mechanisms are not clear.

   Mothers with obesity and/or gestational diabetes have been reported to have obesity-associated gut microbiota. The changes in microbiota could be transmitted to child during vaginal birth. Previously, metagenome sequencing has been succesfully used for comparing the main source of colonization in infants and vertical transmission of gut microbiota and shown that >70% of microbiota is vertically transmitted from the mother to the newborn infant during vaginal delivery.

   In Finland, the rate of C-section has increased from 16-17% to 19.6% of all births. The estimated global average rates are similar, but the C-section rate are expected to increase from the current 21.1% to 28.5%. It is hypnotized that C-section disrupts the vertical transmission of beneficial microbes from the mother to the infant during a critical developmental window. In addition to risk of obesity, C-section increases risk of infectious and chronic diseases such as autoimmune diseases, asthma, and even some cancers.

   Different therapeutic approaches have been proposed and tested for neonatal microbiome restoration in C-section in infants. Intestinal microbes and maternal intestinal strains contribute the most persistent proportion of the neonatal intestinal microbiota after birth, whereas vaginal bacteria and maternal vaginal strains constitute only a small and transient fraction. In two studies, fecal microbiota compositions in infants born by C-section, have succeeded to restore disrupted transmission of intestinal Bacteroides strains by vaginal seeding, while oral administration of the maternal vaginal microbiota to C-section infants had no discernible effect on microbiota composition. In a previous study, fecal transplant from the mother, with a published protocol has been shown to modify the development of infants' gut microbiota successfully and safely.

   As there are evidence, that is possible to modify infants gut microbiota during a critical developmental window, the metabolic consequences and clinical significance of these interventions are unknown. In addition, it is not known what kind of microbiota and from whom would be best for the health of the child in long term.

   The investigators hypothesize that obesity may be a vertically transmitted disease as a newborn child receives obesity-related microbiota from the mother. Furthermore, the source of colonization is a modifiable factor and can be changed by using an early fecal microbiota transplant.
2. STUDY DESIGN AND METHODS

2.1. Recruitment and screening fecal and vaginal samples from the mother

The midwifes and doctors inform potentially participating mothers of the study at the visit and those who are interested to participate are contacted by the study nurse. After informed consent, the mothers are tested for potential contagious diseases as explained below, at the latest 10-14 days before scheduled CS. A fecal sample of 100 g and a blood sample of 15 mL are collected from the mother. The mother divides the feces into the administered sample tubes according to written instructions. Feces for the transplant is collected into an empty tube using a spoon in the cap. The mother informs the research nurse, who delivers the tubes taken for screening to the laboratory as soon as possible, where the transplant is prepared from the fresh sample - this process is completed with a 6 h time frame.

The fresh fecal sample is screened for the presence of parasites and pathogenic viruses and bacteria. An aliquot (0.125 g) of the fresh fecal sample is used to determine the bacterial composition of the sample. Vaginal samples will be obtained during a visit for the assessment of mode of delivery if not already obtained at maternal welfare clinic as a part of routine follow-up.

Blood tests: Complete Blood Count, Erythrocyte sedimentation rate, C-reactive protein, Alanine transaminase, Alkaline phosphatase, Gamma-glutamyl transferase, Albumin, Creatinine, HIV, Hepatitis B, C and E, Treponema pallidum, Human T-cell leukemia virus, CMV ja EBV

Vaginal and perineal screening: Group B Streptococcus, Methicillin-resistant Staphylococcus aureus (MRSA), Extended Spectrum Beta Lactamase (ESBL)

Fecal screening: Salmonella spp., Shigella sp., Campylobacter coli/jejuni, Yersinia enterocolitica, Enterohemorragic E. coli (EHEC), Enteroinvasive E. coli (EIEC), Enterotoxigenic E. coli (ETEC), Vibrio sp., Plesiomonas shigelloides, Clostridium difficile, Cryptosporidium spp., Entamoeba histolytica, Giardia lamblia, Norovirus, Multi drug resistant gram negative bacteria (MDRGN), Vancomycin Resistant Enterococcus (VRE), Listeria monocytogenes, Helicobacter pylori, Sars-CoV-2.

2.2 Fecal micrbiota transplant

Another part of the fresh fecal sample from mother is used as the transplant and for that purpose 1 g of feces is dissolved in 15 mL of isotonic saline and 10% glycerol, homogenized, and the 0.5 mL aliquots of the transplant are immediately frozen and stored at -80 °C.

Fecal transplant from normal weight, healthy female donor (18 to 35 years) from Turku Microbiome Biobank (University of Turku and Turku University Hospital). Donor is tested for potential contagious diseases simultaneously as mother.

2.3 Follow-up in the mother and baby unit

During hospital stay, fecal samples are collected from the first stool of the life and at the age of two to three days. After the first feeding the newborn is followed-up according to the hospital protocols at the rooming-in ward. In previous studies fever has been reported rarely in newborns who have received fecal transplant. Possible adverse events, such as increased peristalsis, diarrhea, vomiting, fever, and rash, are reported to the electronic database of patient records and collected from there by the researchers. Before discharge, the child is weighted and discharge examination is performed by pediatrician or doctor specializing in pediatrics, typically on postnatal day 2.

At the age of 2 days, simultaneously to the screening samples for SCID and metabolic diseases, peripheral blood mononuclear cells (PBMCs) are isolated from capillary blood samples (100µl) drawn from the heel and stored at -140℃. Serum is separated and stored at -80℃. Cells are subjected to analyses, including single cell mRNA sequencing to examine gene expression levels and immunophenotyping by flow cytometry to examine distribution of immune cell types as well as functional properties, including activation and surface receptors. The inflammatory, immunity and obesity related serum components are examined from serum samples (10µl) by high-multiplex Olink or other immunoassays.

2.4 Follow-up after discharge

From the first postnatal week on, the infant is followed in the well-baby clinic according to normal national protocols. As a part of the study, the parents can be in contact with the pediatric emergency department of Oulu University Hospital.

At 3 and 12 months postnatally, parents are asked to fulfill an online questionnaire about child's health and collect and send the fecal samples of the infant and mother to the XXOMNIgeneGUT (DNA genotek, Ontario, Canada) tubes for microbiota analysis and to OMNImetGUT tubes for metabolites and temporarily stored at room temperature before transfer to Turku Microbiome Biobank by mail. At 3 months postnatally, the fecal sample is collected before the second orally given rota virus vaccination, if possible. Fecal samples are not collected during the acute gastrointestinal infection.

DNA from the microbiota samples will be isolated using Chemagic 360 machines and Chemagic Stool 200 H96 kit (PerkinElmer, Turku, Finland). The samples will be sequenced either at the Turku University Hospital, Clinical Microbiology on an Illumina Nextseq 2000 machine or at the Finnish Functional Genomics Centre on an Illumina Novaseq 6000 machine.

Microbiome outcomes:

* 16S next generations sequencing
* Metagenome sequencing and source of colonization
* Microbiome-derived extracellular vesicles: proteome, bacterial 16S
* Microbiota produced metabolites
* Antimicrobial resistance genes

Advanced bioinformatics will be used for microbiome analysis. Source of colonization using metagenome sequencing will be determined as reported earlier.

2.5 Questionnaires

Data are collected on the families' lifestyle, environmental exposures and the health of the study infants and their parents using online questionnaires, enabling monitoring and data query during data collection. Questionnaires are filled by the parents before the birth of the infant and subsequently. Parents are requested to fill in questionnaires on child's nutrition, gastrointestinal function, and care practices in the 3 months, and in the 12 months of age. The questions change as the child grows. Illnesses, medication and use of probiotics and other dietary supplements are reported in the questionnaires. The questionnaires related to nutrition, health and background are mainly similar as in the ongoing HELMi study and Secflor study. To enhance compliance of response rates to the questionnaire, parents receive automatic reminders via email and SMS-messages.

2.6 Patient records

The perinatal data will be obtained from electronic delivery record data concerning newborn's hypoglycemia, follow-up of glucose levels, need for intravenous glucose infusion before discharge from hospital, age at discharge, symptoms of infection, levels of infection parameters and use of antibiotics during hospital stay, will be collected from hospitals patient records. Growth data up to age of three years measured during normal visits to well-baby clinic and vaccination data will be gathered from parents or from well-baby clinics. Use of antibiotics and other medication up to age of three years will be collected via questionnaires and confirmed from Kanta-service with written permission of the parents.

2.7 Power analysis

Resulting from the screening process, a 40% exclusion rate is expected because of group B streptococci (GBS) carrier state 24% of pregnant women in our region and other positive findings in the screening samples. The trial is designed with a planned sample of 150 mothers, allowing the final number of the subjects with an estimated 40% drop-out rate due to screening positivity to be 90 (30 in each intervention group) taking into consideration that it is likely to have drop-outs during the follow-up period. Microbiome data are multidimensional and binary outcomes are not suitable for power analysis.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women age 18-49 years with obesity (prepregnancy BMI ≥ 30 kg/m2) scheduled for elective CS at term, are recruited at 36 weeks of gestation during a visit for the assessment of mode of delivery at Oulu university Hospital, Oulu, Finland.

Exclusion Criteria:

* Use of regular immunosuppressive biological medication, immunodeficiency disorder of mother or other first degree family member of the unborn baby, known or suspected fetal major congenital abnormality, travelling abroad outside European countries or United States within the last three months and antibiotic treatment within 3 months of delivery (excluding the prophylactic cefuroxime (or other in case of allergy) given prior to the elective CS).
* Infant exclusion criteria are preterm birth (birth before 37 weeks of gestation), birth weight below 2500 g, admission to neonatal intensive care unit, need for respiratory support or antibiotic treatment of the newborn before discharge. In case of a suspected infection or newborn screening result for severe combined immunodeficiency (SCID) is out of the normal range, of the newborn the randomization code can be opened.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women.
Enrollment: 150 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Microbial composition profiles in fecal sample | Until 12 months of age
  The difference in microbial composition profiles in fecal sample between the infants in different study groups, specifically diversity and relative abundances of different bacteria phyla and species.
Height in centimeters | 3 years of age
  The difference in growth in height between the infants in different study groups
Height z-score | 3 years of age
  The difference in growth in height between the infants in different study groups
Weight in kilograms | 3 years of age
  The difference in growth in weight in infants the infants in different study groups
Weight-for-length (%) | 3 years of age
  The difference in growth in weight in infants the infants in different study groups

SECONDARY OUTCOMES:
The source of colonization by exclusively shared genes (ESGs) | 3 month of age
  Is the microbiota vertically transmitted from mother or does fecal transplant alter the microbiota measured by ESGs, which are defined as genes that are found in only 2 individuals of all subjects. In the study, the nucleotide sequences of ESGs are required to be 100% identical. As such, ESGs are strong indicators of the transmission of species and genes from one subject to another. If a single species is found in 2 individuals (1 mother, 1 infant) who have ≥1 ESG that belongs to this species, the species is considered a transmitted species.

CONTACTS AND LOCATIONS:
Overall Officials: Terhi Tapiainen, Professor, Principal Investigator — Oulu Univeristy Hospital; Marika Paalanne, MD, PhD, Study Director — Oulu Univeristy Hospital

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.

REFERENCES:
- [Background] Simmonds M, Llewellyn A, Owen CG, Woolacott N. Predicting adult obesity from childhood obesity: a systematic review and meta-analysis. Obes Rev. 2016 Feb;17(2):95-107. doi: 10.1111/obr.12334. Epub 2015 Dec 23. PMID 26696565
- [Background] Korpela K, Renko M, Vanni P, Paalanne N, Salo J, Tejesvi MV, Koivusaari P, Ojaniemi M, Pokka T, Kaukola T, Pirttila AM, Tapiainen T. Microbiome of the first stool and overweight at age 3 years: A prospective cohort study. Pediatr Obes. 2020 Nov;15(11):e12680. doi: 10.1111/ijpo.12680. Epub 2020 Jul 7. PMID 32638554
- [Background] Cho NA, Sales KM, Sampsell K, Wang W, Noye Tuplin EW, Lowry DE, Reimer RA. C-section birth increases offspring obesity risk dependent on maternal diet and obesity status in rats. Obesity (Silver Spring). 2021 Oct;29(10):1664-1675. doi: 10.1002/oby.23258. Epub 2021 Aug 31. PMID 34464518
- [Background] Huh SY, Rifas-Shiman SL, Zera CA, Edwards JW, Oken E, Weiss ST, Gillman MW. Delivery by caesarean section and risk of obesity in preschool age children: a prospective cohort study. Arch Dis Child. 2012 Jul;97(7):610-6. doi: 10.1136/archdischild-2011-301141. Epub 2012 May 23. PMID 22623615
- [Background] Collado MC, Isolauri E, Laitinen K, Salminen S. Distinct composition of gut microbiota during pregnancy in overweight and normal-weight women. Am J Clin Nutr. 2008 Oct;88(4):894-9. doi: 10.1093/ajcn/88.4.894. PMID 18842773
- [Background] Ainonen S, Tejesvi MV, Mahmud MR, Paalanne N, Pokka T, Li W, Nelson KE, Salo J, Renko M, Vanni P, Pirttila AM, Tapiainen T. Antibiotics at birth and later antibiotic courses: effects on gut microbiota. Pediatr Res. 2022 Jan;91(1):154-162. doi: 10.1038/s41390-021-01494-7. Epub 2021 Apr 6. PMID 33824448
- [Background] Betran AP, Ye J, Moller AB, Souza JP, Zhang J. Trends and projections of caesarean section rates: global and regional estimates. BMJ Glob Health. 2021 Jun;6(6):e005671. doi: 10.1136/bmjgh-2021-005671. PMID 34130991
- [Background] Shao Y, Forster SC, Tsaliki E, Vervier K, Strang A, Simpson N, Kumar N, Stares MD, Rodger A, Brocklehurst P, Field N, Lawley TD. Stunted microbiota and opportunistic pathogen colonization in caesarean-section birth. Nature. 2019 Oct;574(7776):117-121. doi: 10.1038/s41586-019-1560-1. Epub 2019 Sep 18. PMID 31534227
- [Background] Podlesny D, Fricke WF. Strain inheritance and neonatal gut microbiota development: A meta-analysis. Int J Med Microbiol. 2021 Apr;311(3):151483. doi: 10.1016/j.ijmm.2021.151483. Epub 2021 Feb 25. PMID 33689953
- [Background] Korpela K, Costea P, Coelho LP, Kandels-Lewis S, Willemsen G, Boomsma DI, Segata N, Bork P. Selective maternal seeding and environment shape the human gut microbiome. Genome Res. 2018 Apr;28(4):561-568. doi: 10.1101/gr.233940.117. Epub 2018 Mar 1. PMID 29496731
- [Background] Decker E, Engelmann G, Findeisen A, Gerner P, Laass M, Ney D, Posovszky C, Hoy L, Hornef MW. Cesarean delivery is associated with celiac disease but not inflammatory bowel disease in children. Pediatrics. 2010 Jun;125(6):e1433-40. doi: 10.1542/peds.2009-2260. Epub 2010 May 17. PMID 20478942
- [Background] Cardwell CR, Stene LC, Joner G, Cinek O, Svensson J, Goldacre MJ, Parslow RC, Pozzilli P, Brigis G, Stoyanov D, Urbonaite B, Sipetic S, Schober E, Ionescu-Tirgoviste C, Devoti G, de Beaufort CE, Buschard K, Patterson CC. Caesarean section is associated with an increased risk of childhood-onset type 1 diabetes mellitus: a meta-analysis of observational studies. Diabetologia. 2008 May;51(5):726-35. doi: 10.1007/s00125-008-0941-z. Epub 2008 Feb 22. PMID 18292986
- [Background] Keag OE, Norman JE, Stock SJ. Long-term risks and benefits associated with cesarean delivery for mother, baby, and subsequent pregnancies: Systematic review and meta-analysis. PLoS Med. 2018 Jan 23;15(1):e1002494. doi: 10.1371/journal.pmed.1002494. eCollection 2018 Jan. PMID 29360829
- [Background] Stokholm J, Thorsen J, Blaser MJ, Rasmussen MA, Hjelmso M, Shah S, Christensen ED, Chawes BL, Bonnelykke K, Brix S, Mortensen MS, Brejnrod A, Vestergaard G, Trivedi U, Sorensen SJ, Bisgaard H. Delivery mode and gut microbial changes correlate with an increased risk of childhood asthma. Sci Transl Med. 2020 Nov 11;12(569):eaax9929. doi: 10.1126/scitranslmed.aax9929. PMID 33177184
- [Background] Ferretti P, Pasolli E, Tett A, Asnicar F, Gorfer V, Fedi S, Armanini F, Truong DT, Manara S, Zolfo M, Beghini F, Bertorelli R, De Sanctis V, Bariletti I, Canto R, Clementi R, Cologna M, Crifo T, Cusumano G, Gottardi S, Innamorati C, Mase C, Postai D, Savoi D, Duranti S, Lugli GA, Mancabelli L, Turroni F, Ferrario C, Milani C, Mangifesta M, Anzalone R, Viappiani A, Yassour M, Vlamakis H, Xavier R, Collado CM, Koren O, Tateo S, Soffiati M, Pedrotti A, Ventura M, Huttenhower C, Bork P, Segata N. Mother-to-Infant Microbial Transmission from Different Body Sites Shapes the Developing Infant Gut Microbiome. Cell Host Microbe. 2018 Jul 11;24(1):133-145.e5. doi: 10.1016/j.chom.2018.06.005. PMID 30001516
- [Background] Mitchell CM, Mazzoni C, Hogstrom L, Bryant A, Bergerat A, Cher A, Pochan S, Herman P, Carrigan M, Sharp K, Huttenhower C, Lander ES, Vlamakis H, Xavier RJ, Yassour M. Delivery Mode Affects Stability of Early Infant Gut Microbiota. Cell Rep Med. 2020 Dec 22;1(9):100156. doi: 10.1016/j.xcrm.2020.100156. eCollection 2020 Dec 22. PMID 33377127
- [Background] Dominguez-Bello MG, De Jesus-Laboy KM, Shen N, Cox LM, Amir A, Gonzalez A, Bokulich NA, Song SJ, Hoashi M, Rivera-Vinas JI, Mendez K, Knight R, Clemente JC. Partial restoration of the microbiota of cesarean-born infants via vaginal microbial transfer. Nat Med. 2016 Mar;22(3):250-3. doi: 10.1038/nm.4039. Epub 2016 Feb 1. PMID 26828196
- [Background] Song SJ, Wang J, Martino C, Jiang L, Thompson WK, Shenhav L, McDonald D, Marotz C, Harris PR, Hernandez CD, Henderson N, Ackley E, Nardella D, Gillihan C, Montacuti V, Schweizer W, Jay M, Combellick J, Sun H, Garcia-Mantrana I, Gil Raga F, Collado MC, Rivera-Vinas JI, Campos-Rivera M, Ruiz-Calderon JF, Knight R, Dominguez-Bello MG. Naturalization of the microbiota developmental trajectory of Cesarean-born neonates after vaginal seeding. Med. 2021 Aug 13;2(8):951-964.e5. doi: 10.1016/j.medj.2021.05.003. Epub 2021 Jun 17. PMID 35590169
- [Background] Wilson BC, Butler EM, Grigg CP, Derraik JGB, Chiavaroli V, Walker N, Thampi S, Creagh C, Reynolds AJ, Vatanen T, O'Sullivan JM, Cutfield WS. Oral administration of maternal vaginal microbes at birth to restore gut microbiome development in infants born by caesarean section: A pilot randomised placebo-controlled trial. EBioMedicine. 2021 Jul;69:103443. doi: 10.1016/j.ebiom.2021.103443. Epub 2021 Jun 27. PMID 34186487
- [Background] Helve O, Dikareva E, Stefanovic V, Kolho KL, Salonen A, de Vos WM, Andersson S. Protocol for oral transplantation of maternal fecal microbiota to newborn infants born by cesarean section. STAR Protoc. 2021 Jan 15;2(1):100271. doi: 10.1016/j.xpro.2020.100271. eCollection 2021 Mar 19. PMID 33511356
- [Background] Carpen N, Brodin P, de Vos WM, Salonen A, Kolho KL, Andersson S, Helve O. Transplantation of maternal intestinal flora to the newborn after elective cesarean section (SECFLOR): study protocol for a double blinded randomized controlled trial. BMC Pediatr. 2022 Sep 29;22(1):565. doi: 10.1186/s12887-022-03609-3. PMID 36175995
- [Background] Korpela K, Dikareva E, Hanski E, Kolho KL, de Vos WM, Salonen A. Cohort profile: Finnish Health and Early Life Microbiota (HELMi) longitudinal birth cohort. BMJ Open. 2019 Jun 27;9(6):e028500. doi: 10.1136/bmjopen-2018-028500. PMID 31253623
- [Background] Saari A, Sankilampi U, Hannila ML, Kiviniemi V, Kesseli K, Dunkel L. New Finnish growth references for children and adolescents aged 0 to 20 years: Length/height-for-age, weight-for-length/height, and body mass index-for-age. Ann Med. 2011 May;43(3):235-48. doi: 10.3109/07853890.2010.515603. Epub 2010 Sep 21. PMID 20854213
- [Background] Li W, Tapiainen T, Brinkac L, Lorenzi HA, Moncera K, Tejesvi MV, Salo J, Nelson KE. Vertical Transmission of Gut Microbiome and Antimicrobial Resistance Genes in Infants Exposed to Antibiotics at Birth. J Infect Dis. 2021 Oct 13;224(7):1236-1246. doi: 10.1093/infdis/jiaa155. PMID 32239170